CLINICAL TRIAL: NCT04733079
Title: Treat-to-target by Email During Urate-lowering Therapy in Gout
Acronym: GOUTEmail
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180167
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Gout; Inflammatory Rheumatism; Hyperuricemia; Posology Adjustment
Keywords: Treat-to-target; Gout; Tophus; Urate crystals; Urate-lowering therapy; Febuxostat; Allopurinol; Therapeutic strategy; Electronic messaging; Therapeutic compliance
MeSH Terms: conditions — Gout; Rheumatic Fever; Hyperuricemia; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-mail follow-up group (Experimental): Email-led treat-to-target strategy with regular adaptation of ULT via electronic messaging
  Interventions: Other: Cleanweb electronic messaging ePro
- Usual follow-up group (Active Comparator): Adaptation and follow-up of ULT according to referring physician's habits
  Interventions: Other: Usual follow-up

INTERVENTIONS:
Other: Cleanweb electronic messaging ePro — Patient and their medecin will communicate regulary via Cleanweb electronic messaging ePro to adapt the posology of THU untill the target urecemia is reached
  Arms: E-mail follow-up group
Other: Usual follow-up — Adaptation and follow-up of ULT according to referring physician's habits
  Arms: Usual follow-up group

SUMMARY:
Gout is secondary to urate crystal deposition after chronic elevation of serum urate level (SUL). Long-term lowering SUL below 360 µmol/L allows dissolution of deposited crystals and disease cure. There is currently a paradoxical observation: while urate-lowering therapy (ULT) is available and efficient there is an increase of gout prevalence and severity. The apparent failure of ULT in gout management is due to several causes including unadjusted dosage, no SUL verification, irregular follow-up and low treatment compliance.

In contrast, a nurse-led treat-to-target (T2T) strategy with regular adaptations of ULT until reaching SUL target allows gout cure in more than 90% of patients. We hypothesize that an electronic messaging-led T2T strategy will allow obtaining similar results.

The aim of this study is to demonstrate that email-led T2T strategy during ULT is superior to usual care.

DETAILED DESCRIPTION:
The study will include 204 gouty patients without ULT or with ineffective ULT. This is a multicenter and randomized study (e-mail follow-up vs usual follow-up groups).

This study will include the following visits:

* Selection/inclusion visit (V0):

  * If available biological data (leucocyte count, hemoglobin level, creatininemia and estimated glomerular filtration rate (eGFR), SUL) were assessed during the last month, , included patient will be randomized at the end of the consultation to follow either an email-led T2T strategy or usual ULT care.
  * In the absence of biological results, the patient will be reviewed within the month with blood analysis and then randomized.
* Follow-up visits: consultations will be carried out according to the usual care of the referring physician.
* Visit M12 end of research: clinical evaluation of gout, demographic characteristics, medication, type and dose of ULT, blood analysis (serum creatinine level, eGFR, SUL).

The study ends after the M12 consultation. The total duration of participation in the study is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years old
* Gout confirmed by identification of urate crystals by joint fluid or tophus analysis or by ultrasound of the affected joint or
* Gout according to Nijmegen criteria (presence of a score ≥ 8/13) depending on the following items:

Man (2 pts) Previous crisis (2 pts) Involvement of first metatarsophalangeal joint (MTP1) (2.5 pts) Maximum pain within 24 hours (0.5pt) Redness (1 pt) HTA or cardiovascular disease (1.5 pts) SUL > 360 μmol/l during the crisis (3.5 pts)

* Patients without ULT or with an ineffective ULT defined by an SUL > 360 μmol/l in intercritical pahse
* Patients who routinely use e-mail

Exclusion Criteria:

* Participating in another trial including the administration of a drug
* Patients treated with azathioprine
* Patients intolerant to hypouricemic treatments
* Unable to use the internet
* Difficulty understanding French
* Illiteracy
* Pregnant womenor breastfeeding mothers (see PHC article L.1121-5)
* Persons deprived of liberty by judicial or administrative decision, persons receiving psychiatric care under Sections L. 3212-1 and L. 3213-1 and persons admitted to a health or social institution for purposes other than research (see CSP Article L.1121-6)
* Major persons subject to a measure of legal protection or unseeding to express consent (see PHC Article L.1121-8)
* Persons not affiliated to a social security plan or beneficiaries of such a plan (see PHC Article L.1121-8-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with target SUL (<360 μmol /L or <300 μmol /L in tophaceous gout) | Month 12

SECONDARY OUTCOMES:
Average dose of ULT (allopurinol and febuxostat) | Month 12

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital LARIBOISIERE - Rhumatologie, Paris
  - Rhumathology department, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No